CLINICAL TRIAL: NCT03124368
Title: A Phase 2a Proof-of-Mechanism, Open-Label Study to Determine the Effect of ACH-0144471 on C3 Levels in Participants With Low C3 Levels Due to Either C3 Glomerulopathy (C3G) or Immune-Complex Membranoproliferative Glomerulonephritis (IC-MPGN)
Brief Title: A Proof-of-Mechanism Study to Determine the Effect of Danicopan on C3 Levels in Participants With C3G or IC-MPGN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: ACH471-201; 2016-003525-42 (EudraCT Number)
Record Dates: First submitted 2017-04-12; First posted 2017-04-21 (Actual); Results first posted 2021-07-13 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: C3 Glomerulonephritis; Dense Deposit Disease; C3 Glomerulopathy; Immune Complex Mediated Membranoproliferative Glomerulonephritis; Membranoproliferative Glomerulonephritis Types I, II, and III
Keywords: factor D; FD; alternative pathway; complement mediated disease; idiopathic MPGN; MPGN Type I; MPGN Type II; MPGN Type III; Primary MPGN; MCGN; Mesangiocapillary Glomerulonephritis; C3 Glomerulopathy; C3G; Membranoproliferative Glomerulonephritis; C3GN; Dense Deposit Disease; DDD
MeSH Terms: conditions — Glomerulonephritis, Membranoproliferative | interventions — danicopan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: Danicopan 100 mg TID (Sentinel) (Experimental): All participants received 100 milligrams (mg) of danicopan three times per day (TID) during the Treatment Period.
  Interventions: Drug: Danicopan
- Group 2: Danicopan up to 200 mg TID (Experimental): All participants received not more than 200 mg of danicopan TID depending on the available safety, pharmacokinetic, and pharmacodynamic data from Group 1 (Sentinel) during the Treatment Period.
  Interventions: Drug: Danicopan

INTERVENTIONS:
Drug: Danicopan — Participants received study drug for 14 days (Treatment Period), followed by a taper over the next 7 days (Taper Period).
  Other Names: ACH-4471; ACH4471; 4471; ACH-0144471; ALXN2040

SUMMARY:
The primary objective of this study was to determine whether ACH-0144471 (also known as danicopan and ALXN2040) increases blood C3 complement protein (C3) levels in participants with low C3 levels due to either C3G or IC-MPGN.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have had clinical diagnosis of C3G (C3 glomerulonephritis or dense deposit disease, the 2 types of C3G) or idiopathic IC-MPGN by renal biopsy for at least 3 months prior to dosing, with the pathologic diagnosis verified by a review of the renal biopsy by the study central pathologist
* C3 must have been <50% of the lower limit of normal
* C4 complement protein (C4) must have been >90% of the lower limit of normal
* Must have been willing to comply with study-specific vaccination requirements for Haemophilus influenzae, Streptococcus pneumoniae, and Neisseria meningitidis strains A, C, W, and Y
* Negative pregnancy test for females prior to dosing and throughout the study

Key Exclusion Criteria:

* History of a major organ transplant (for example, heart, lung, kidney, liver) or hematopoietic stem cell/marrow transplant. Individuals receiving renal replacement therapy were also excluded
* Evidence of monoclonal gammopathy of unclear significance, infections, malignancy, autoimmune diseases, or other conditions to which C3G or IC-MPGN may have been secondary
* Estimated glomerular filtration rate (using Modification of Diet in Renal Disease equation) <45 milliliters/minute/1.73 square meters at the time of Screening or at any time over the preceding 4 weeks
* Receipt of eculizumab at any dose or interval within the past 75 days prior to dosing
* Use of tacrolimus or cyclosporine within 2 weeks of the first dose of danicopan
* History of febrile illness, a body temperature >38°Celsius, or other evidence of a clinically significant active infection, within 14 days prior to study drug administration
* History of meningococcal infection, or a first-degree relative or household contact with a history of meningococcal infection
* Females who were pregnant, nursing, or planning to become pregnant during the study or within 90 days of study drug administration or participants with a female partner who was pregnant, nursing, or planning to become pregnant during the study or within 90 days of study drug administration

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-01-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Clinical Trial Site, Melbourne, Australia
- Clinical Trial Site, Antwerp, Belgium
- Clinical Trial Site, Leiden, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 5 study centers total in Australia, Belgium, and The Netherlands. Only 3 study centers, 1 in each country, treated participants.
Groups:
- Group 1: Danicopan 100 mg TID (Sentinel): Participants received 100 milligrams (mg) of danicopan three times daily (TID) during the Treatment Period.
- Group 2: Danicopan up to 200 mg TID: Participants received not more than 200 mg of danicopan TID during the Treatment Period.
Period: Overall Study
Arm/Group | Group 1: Danicopan 100 mg TID (Sentinel) | Group 2: Danicopan up to 200 mg TID
Started | 2 | 4
Received at Least 1 Dose of Study Drug | 2 | 4
Completed | 2 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of danicopan.
Groups:
- Group 1: Danicopan 100 mg TID (Sentinel): Participants received 100 mg of danicopan TID during the Treatment Period.
- Total: Total of all reporting groups
Arm/Group | Group 1: Danicopan 100 mg TID (Sentinel) | Group 2: Danicopan up to 200 mg TID | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.50 (7.85) | 30.00 (12.68) | 28.50 (10.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 3 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline In Serum C3 Complement Protein (C3) Levels On Day 15
Description: Serum C3 levels were measured by conventional Roche immunoturbidimetric assay method.
  Change from Baseline = Serum C3 levels on Day 15 - Baseline Serum C3 levels
Time Frame: Baseline, Day 15
Population: All participants who received at least 1 dose of danicopan and who had a baseline measurement and at least 1 measurement during the treatment period.
Measure: Mean (Standard Deviation); unit: g/L
Groups:
- Total: All participants who received at least 1 dose of danicopan.
Arm/Group | Group 1: Danicopan 100 mg TID (Sentinel) | Group 2: Danicopan up to 200 mg TID | Total
Number analyzed (Participants) | 2 | 4 | 6
g/L
  Baseline | 0.32 (0.060) | 0.56 (0.230) | 0.48 (0.220)
  Day 15 | 0.35 (0.060) | 0.70 (0.350) | 0.58 (0.330)
  Change from Baseline | 0.03 (0.000) | 0.14 (0.140) | 0.11 (0.120)

2. Primary Outcome: Change From Baseline In Plasma Intact C3 Level On Day 15
Description: Plasma Intact C3 level were measured by a novel multiplex assay method. Change from Baseline = Plasma Intact C3 levels on Day 15 - Baseline Plasma Intact C3 levels
Time Frame: Baseline, Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Group 1: Danicopan 100 mg TID (Sentinel) | Group 2: Danicopan up to 200 mg TID | Total
Number analyzed (Participants) | 2 | 4 | 6
μg/mL
  Baseline | 39.50 (0.710) | 58.25 (47.910) | 52.00 (38.360)
  Day 15 | 54.30 (17.390) | 33.50 (9.040) | 40.43 (15.000)
  Change from Baseline | 14.80 (18.100) | -24.75 (50.970) | -11.57 (45.180)

3. Secondary Outcome: Change From Baseline In Total Complement Classical Pathway (CP) Activity On Day 14
Description: CP activity was measured in serum by the DiaSorin Complement Activation Enzyme (CAE) functional immunoassay method, which measures terminal complement complex formation following activation. Results are expressed in CAE units which are calculated relative to previously established CAE activity of a positive control serum.
  Change from Baseline = Total Complement CP Activity on Day 14 - Baseline Total Complement CP Activity
Time Frame: Baseline, Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CAE unit
Arm/Group | Group 1: Danicopan 100 mg TID (Sentinel) | Group 2: Danicopan up to 200 mg TID | Total
Number analyzed (Participants) | 2 | 4 | 6
CAE unit
  Baseline | 31.00 (21.210) | 91.00 (41.370) | 71.00 (45.570)
  Day 14 | 41.50 (23.330) | 96.75 (23.680) | 78.33 (35.490)
  Change from Baseline | 10.50 (2.120) | 5.75 (34.250) | 7.33 (26.660)

4. Secondary Outcome: Change From Baseline In Total Complement Alternative Pathway (AP) Functional Activity (AP Wieslab) On Day 15
Description: AP functional activity was measured in serum by the Wieslab functional immunoassay method, which measures terminal complement complex (TCC) formation following AP-specific activation. Results are expressed as percent TCC production relative to a positive control serum.
  Change from Baseline = Total Complement AP Functional Activity on Day 15 - Baseline Total Complement AP Functional Activity
Time Frame: Baseline, Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of activity
Arm/Group | Group 1: Danicopan 100 mg TID (Sentinel) | Group 2: Danicopan up to 200 mg TID | Total
Number analyzed (Participants) | 2 | 4 | 6
percentage of activity
  Baseline | 8.350 (10.508) | 31.073 (19.779) | 23.498 (19.862)
  Day 15 | 1.635 (2.3122) | 0.993 (1.1101) | 1.207 (1.3852)
  Change from Baseline | -6.715 (8.1954) | -30.08 (19.176) | -22.29 (19.484)

5. Secondary Outcome: Time To Achieving Peak Serum C3 Levels
Description: Serial serum samples were collected on Days 1, 7, and 14.
Time Frame: From The First Day Of Dosing through Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group 1: Danicopan 100 mg TID (Sentinel) | Group 2: Danicopan up to 200 mg TID | Total
Number analyzed (Participants) | 2 | 4 | 6
days | 2.5 (2.12) | 10.5 (4.43) | 7.8 (5.46)

6. Secondary Outcome: Number Of Participants With Serious Adverse Events (SAEs), Grade 3 And Grade 4 Treatment-emergent Adverse Events (TEAEs), And Adverse Events (AEs) Leading To Discontinuation
Description: An AE was as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An SAE was an AE that met at least 1 of the following criteria: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization for the AE, persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug), important medical event or reaction. The intensity of an AE was graded according to the Common Terminology Criteria for Adverse Events (CTCAE) Adverse Event Severity Grading Table. A summary of SAEs and other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Up to Day 49
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Danicopan 100 mg TID (Sentinel) | Group 2: Danicopan up to 200 mg TID | Total
Number analyzed (Participants) | 2 | 4 | 6
Participants
  TEAEs | 2 | 3 | 5
  SAEs | 0 | 1 | 1
  TEAEs ≥Grade 3 | 0 | 0 | 0
  TEAEs leading to discontinuation | 0 | 0 | 0

7. Secondary Outcome: Pharmacokinetics (PK): Area Under The Plasma Concentration-time Curve From Time Of Administration To 8 Hours Postdose (AUC0-8)
Description: Serial blood samples were collected at 0, 1, 1.5, 2, 2.5, 3, 4, 6, and 8 hours post-dose on Days 1 and 7.
Time Frame: Days 1 and 7
Population: All participants receiving at least 1 dose of danicopan who had a baseline measurement and at least 1 measurement during the treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Group 1: Danicopan 100 mg TID: Participants received 100 mg of danicopan TID during the Treatment Period.
- Group 2: Danicopan 150 mg TID: Participants received 150 mg of danicopan TID during the Treatment Period.
- Group 2: Danicopan 200 mg TID: Participants received 200 mg of danicopan TID during the Treatment Period.
Arm/Group | Group 1: Danicopan 100 mg TID | Group 2: Danicopan 150 mg TID | Group 2: Danicopan 200 mg TID
Number analyzed (Participants) | 2 | 1 | 3
h*ng/mL
  Day 1 | 871 (38.1) | 2060 | 1640 (42.8)
  Day 7 | 1120 (44.4) | 2470 | 1760 (24.2)

8. Secondary Outcome: PK: Maximum Plasma Concentration (Cmax)
Description: Serial blood samples were collected at 0, 1, 1.5, 2, 2.5, 3, 4, 6, and 8 hours post-dose on Days 1 and 7.
Time Frame: Days 1 and 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group 1: Danicopan 100 mg TID | Group 2: Danicopan 150 mg TID | Group 2: Danicopan 200 mg TID
Number analyzed (Participants) | 2 | 1 | 3
ng/mL
  Day 1 | 199 (6.75) | 563 | 427 (46.3)
  Day 7 | 270 (41.2) | 579 | 385 (39.1)

9. Secondary Outcome: PK: Time To Maximum Concentration (Tmax)
Description: Serial blood samples were collected at 0, 1, 1.5, 2, 2.5, 3, 4, 6, and 8 hours post-dose on Days 1 and 7.
Time Frame: Days 1 and 7
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1: Danicopan 100 mg TID | Group 2: Danicopan 150 mg TID | Group 2: Danicopan 200 mg TID
Number analyzed (Participants) | 2 | 1 | 3
hours
  Day 1 | 1.00 [1.00 to 1.00] | 2.50 [2.50 to 2.50] | 2.00 [1.50 to 2.00]
  Day 7 | 2.75 [1.50 to 4.00] | 2.50 [2.50 to 2.50] | 1.50 [1.00 to 4.00]

10. Secondary Outcome: Change From Baseline In Bb Fragment Of Complement Factor B (Bb) At Day 15
Description: Plasma Bb was measured by enzyme-linked immunosorbent assay (ELISA).
  Change from Baseline = Complement Bb on Day 15 - Baseline
Time Frame: Baseline, Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Group 1: Danicopan 100 mg TID (Sentinel) | Group 2: Danicopan up to 200 mg TID | Total
Number analyzed (Participants) | 2 | 4 | 6
µg/mL
  Baseline | 1.789 (1.2116) | 1.229 (0.4729) | 1.416 (0.7152)
  Day 15 | 1.511 (0.9781) | 0.622 (0.3349) | 0.918 (0.6854)
  Change from baseline | -0.278 (0.2335) | -0.607 (0.1790) | -0.497 (0.2430)

11. Secondary Outcome: Change From Baseline In Soluble Terminal Complement Complex (sC5b-9) At Day 15
Description: Plasma sC5b-9 was measured by ELISA.
  Change from Baseline = sC5b-9 on Day 15 - Baseline sC5b-9
Time Frame: Baseline, Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1: Danicopan 100 mg TID (Sentinel) | Group 2: Danicopan up to 200 mg TID | Total
Number analyzed (Participants) | 2 | 4 | 6
ng/mL
  Baseline | 1002.0 (684.4794) | 613.750 (225.2397) | 743.167 (405.3874)
  Day 15 | 1105.5 (622.9611) | 563.850 (302.4446) | 744.400 (459.0596)
  Change from Baseline | 103.500 (61.5183) | -49.900 (237.1917) | 1.233 (201.9602)

ADVERSE EVENTS:
Time Frame: After the first dose of study medication (following Day 0) through the follow-up visit at Day 49.
Description: [Not specified]
Arm/Group | Group 1: Danicopan 100 mg TID (Sentinel) | Group 2: Danicopan up to 200 mg TID
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/4
Other Adverse Events (participants affected / at risk) | 2/2 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Danicopan 100 mg TID (Sentinel) (N=2) | Group 2: Danicopan up to 200 mg TID (N=4)
Presyncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Danicopan 100 mg TID (Sentinel) (N=2) | Group 2: Danicopan up to 200 mg TID (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Crepitations (General disorders) | 0 | 1
Prerenal failure (Renal and urinary disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The sample size of the study was based on very limited clinical cases of C3G and IC-MPGN and the exploratory nature of this study to evaluate the effectiveness of danicopan.

Plasma intact C3 values should be regarded with caution. Plasma intact C3 values were generated using a new multiplex assay method with limited historical experience, and internal studies have suggested this new assay is subject to unexplained experimental variation arising during sample preparation and handling.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT03124368/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT03124368/SAP_001.pdf